CLINICAL TRIAL: NCT05969353
Title: Assessing the Effectiveness of BFA as a Non-pharmacologic Pain Management Intervention: A Randomised Sham Controlled Study in Participants Who Hospitalized in Department of Internal Medicine
Brief Title: Assessing the Effectiveness of BFA as a Non-pharmacologic Pain Management Intervention: A Randomised Sham Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, shira.ginsberg, MD, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 062-23 BNZ
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Assessing the Effectiveness of BFA as a Non-pharmacologic Pain Management Intervention: A Randomised Sham Controlled Study

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham controlled arm (Sham Comparator)
  Interventions: Other: accupunture
- battlefield acupunture (Active Comparator)
  Interventions: Other: accupunture

INTERVENTIONS:
Other: accupunture — BFA

SUMMARY:
This is a randomized sham controlled study that will include patients hospitalized in the internal medicine department and the orthopedics department at Bnei Zion Hospital presenting with pain from various sources with an NRS level equal to or above 4.

DETAILED DESCRIPTION:
All patients will complete pain assessment according NSR and ESAS after treatment ( SHAM or BFA) one hour before and every 24 hours until discharge.

If there was no sufficient improvement in pain within 24 hours (decrease of 1.5 points or more in NRS) - additional acupuncture will be performed in the contralateral ear and repeated assessments as above.

ELIGIBILITY:
Inclusion Criteria:

-1.Pain of skeletal muscle origin (Musculoskeletal MSK)/rheumatological/orthopedic syndromes 2.Visual Analog Score (VAS) grade 4 or higher before receiving the treatment.

3.Eligible to participate in the study according to the assessment of the investigator

Exclusion Criteria:

1. Pain syndromes of non-muscular bony/rheumatological/orthopedic origin
2. Planned an MRI next week
3. An infectious process in the ear planned for acupuncture or a history of sensitivity to metal
4. have any participant condition that ' according to the Investigator ' could interfere with the conduct of the trial -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-23 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
efficacy of BFA | two years
  Evaluating the analgesic efficacy of BFA in addition to the standard treatment for pain - Standard of care (SOC) to reduce pain in patients hospitalized in the internal and orthopedic department who experience pain of moderate intensity and above compared to SHAM BFA.

CONTACTS AND LOCATIONS:
Overall Officials: shira ginsberg, MD, Principal Investigator — BnaiZion MC
Locations (1):
- BnaiZion MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided